CLINICAL TRIAL: NCT03547310
Title: PlayBionic: Interactive Mobile Training App After Nerve Transfer or Amputation of the Upper Extremity
Brief Title: PlayBionic: Interactive Mobile Training App
Acronym: PlayBionic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Cosima Prahm, MSc, BA, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1193/2017
Record Dates: First submitted 2018-04-24; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Rehabilitation
Keywords: EMG; Prosthesis control; Neuromuscular rehabilitation; Games for health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MyoBeatz (Experimental): The intervention consists of playing with the smartphone training program using the muscle signals picked up by surface electrodes. The study will run over a period of 5 weeks, with participants playing with the training program at home for 4 weeks.
  Interventions: Behavioral: MyoBeatz

INTERVENTIONS:
Behavioral: MyoBeatz — Training of the patient's muscle coordination, strength and ability to separately contract muscles, while holding up patient motivation. The patient is expected to follow a protocol of 4 weeks of training.

SUMMARY:
Often prosthesis users abandon their devices due to difficulties in prosthesis control and lack of motivation to train. To properly control a prosthesis, amputation patients must learn how to activate, isolate and sustain nerve signals to the muscles left at the stump. Results of clinical validations show that game-based training leads to an improvement in clinical parameters for prosthesis control and patient engagement.

DETAILED DESCRIPTION:
Relevance:

Many users of a myoelectric arm prosthesis do not use their device because they find it too difficult to control the prosthesis. This may be due to the fact that patients cannot contract their muscles in the residual limb in a sufficiently controlled manner. Exactly this circumstance is trained during the physiotherapy with the patients. But at home many patients lack the motivation to continue the exercises from physiotherapy. Mobile games on the smartphone can provide patients with long-term motivation to continue the repetitive exercises that prepare the muscles for controlling a prosthesis at home.

Aim:

The aim of this study is to support patients in training at home with a game on their smartphone. This should increase motivation and improve the ability to control a prosthesis efficiently.

Design:

The Smartphone App is a rhythmic, music-based game consisting of different game modes. It has not only a display for real-time bio-feedback, but also many other audiovisually motivating incentives to continue playing the game. Similar to the classical control of a commercial prosthesis, the muscle signals are measured by two surface electrodes and, in this case, transferred to the app instead of the prosthesis. With these 2 electrodes the game is controlled. Test persons receive feedback on their performance through the constantly displayed bio-feedback, but also through high scores of the various levels and user statistics. By testing the muscle coordination twice a week, the neuromuscular improvements in the control of the game can be monitored.

Method/Procedure:

Eight transradially (below the elbow) amputated patients participate in this study. The intervention consists of playing with the smartphone training program using the muscle signals picked up by surface electrodes. The study will run over a period of 5 weeks, with participants playing with the training program at home for 4 weeks. The program should be used 5 times per week, therefore the intervention takes place 20 times in total. In the 5th week the final assessment, a final evaluation and the return of the devices take place. All usage data, such as starting and exiting the program and the duration of use, are recorded by the program itself and treated anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Transradial amputees are included in the study.

Exclusion Criteria:

* Exclusion criterion is the inappropriate handling of the Android tablet or the computer ,as well as cyber sickness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Voluntary Contraction | 10 minutes
  Testing the patients voluntary myoelectric (EMG) contraction strength, given in millivolt (mV).
  This assessment is used as a calibration of the voltage detected by the electrodes. Participants are asked to maximally contract one muscle and to hold this contraction for 1.3 seconds, of which only the last second is taken for calculating the activation baseline.
Precision Control | 30 minutes
  Testing the patient's ability to precisely control their muscle contraction, given in percentage of target deviation.
  The Assessment of Precision Control evaluates the participant's fine EMG control accuracy. The range of this test was adapted based on the outcome of the MVC test. The participant is asked to reach 30 randomly preselected activation levels in the range of 10-90% of maximum voluntary contraction, and sustain them for 300 milliseconds each. The required level of activation is indicated by a triangular mark on the EMG bar. A total of 30 marks (3 trials consisting of 10 levels) are performed. The percentile deviation from the mark is taken as outcome measure.
Endurance Control | 15 minutes
  The Assessment of Endurance Control assesses muscle coordination and muscle fatigue while the participants used their EMG signals to closely follow a sine curve o 1/4 hertz on the screen until they feel fatigued. The estimated force needed to reach the peaks of the sine curve corresponds to 60% maximum voluntary contraction. Electrode activation needs to be separate to reach the peaks of the sine curve. The minimum time to be reached in this test is 5 minutes. The outcome measure is the EMG signal deviation from the desired sine curve, given as correlation r².

SECONDARY OUTCOMES:
Phantom limb pain | At the beginning and at the end of the study (after 4 weeks)
  Evaluation if the patient's phantom limb pain has been alleviated during or after the intervention. A questionnaire will be given that includes questions from the MPI - German version of the Multidimensional Pain Inventory. Three parts of the inventory, comprised of 12 scales, examine the impact of pain on the patients' lives, the responses of others to the patients' communications of pain, and the extent to which patients participate in common daily activities. The outcome measure is a number that will represent the pain felt by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Aszmann, Prof., Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, CD Laboratory for Restoration of Extremity Function, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prahm C, Vujaklija I, Kayali F, Purgathofer P, Aszmann OC. Game-Based Rehabilitation for Myoelectric Prosthesis Control. JMIR Serious Games. 2017 Feb 9;5(1):e3. doi: 10.2196/games.6026. PMID 28183689